CLINICAL TRIAL: NCT00570752
Title: A 12-Week, Randomized, Semi Double-Blinded Study Evaluating the Effects of Daily Oral High-Dose Atorvastatin or BMS-582949 on Atherosclerotic Plaque Inflammation as Determined by FDG-PET in High Risk Atherosclerotic Patients
Brief Title: Efficacy Study of p38 Kinase Inhibitor to Treat Patients With Atherosclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IM119-014
Record Dates: First submitted 2007-12-10; First posted 2007-12-11 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-11

CONDITIONS: Vascular Diseases
MeSH Terms: conditions — Vascular Diseases | interventions — 4-(5-(cyclopropylcarbamoyl)-2-methylphenylamino)-5-methyl-N-propylpyrrolo(1,2-f)(1,2,4)triazine-6-carboxamide; Atorvastatin; Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo + background low to moderate dose statin (Active Comparator): Placebo + background low to moderate dose statin Tablets, Oral, 0 mg, once daily, for 12 weeks
  Interventions: Other: Placebo; Drug: Statin
- BMS-582949 + Background low to moderate dose statin (Experimental): BMS-582949 + Background low to moderate dose statin Tablets, Oral, 100 mg, once daily for 12 weeks
  Interventions: Drug: BMS-582949; Drug: Statin
- Atorvastatin (Active Comparator): Atorvastatin Tablets, oral, 80 mg once daily for 12 weeks
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Other: Placebo
  Arms: Placebo + background low to moderate dose statin
Drug: BMS-582949
  Arms: BMS-582949 + Background low to moderate dose statin
Drug: Atorvastatin
  Arms: Atorvastatin
Drug: Statin
  Arms: BMS-582949 + Background low to moderate dose statin; Placebo + background low to moderate dose statin

SUMMARY:
The purpose of the study is to determine whether a p38 kinase inhibitor reduces inflammation in atherosclerotic plaque

ELIGIBILITY:
Inclusion Criteria:

* History of documented atherosclerosis
* LDL between 70 and 130 mg/dL
* Patients receiving stable low- to moderate-dose statin
* BMI 18-37 kg/m²
* Must be able to swallow tablets
* Must be able to medically tolerate the procedures, contrast medium, and medications involved

Exclusion Criteria:

* Statin intolerance
* Renal impairment (serum creatinine > 1.5 mg/dL)
* History of chronic viral hepatitis or other liver dysfunction
* Major infection requiring hospitalization or receipt of IV antibiotics due to an infection within 2 months prior to initiation of study treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2008-12; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
FDG-PET signal of the carotid and/or ascending aorta | at 4 and 12 weeks

SECONDARY OUTCOMES:
Inflammatory and thrombotic biomarkers | will be measured throughout the 12 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (17):
- United States (17):
  - Southeast Clinical Research, Llc, Chiefland, Florida
  - Jacksonville Center For Clinical Research - Univ Campus, Jacksonville, Florida
  - Florida Cardiovascular Institute, Tampa, Florida
  - Phillip D. Toth, Md, Indianapolis, Indiana
  - L-Marc Research Center, Louisville, Kentucky
  - Commonwealth Biomedical Research, Llc, Madisonville, Kentucky
  - Mgh Cardiac Mr Pet Ct Program, Boston, Massachusetts
  - Troy Internal Medince Pc/Research, Troy, Michigan
  - Radiant Research, Inc., Edina, Minnesota
  - Mount Sinai School Of Medicine Imaging Science Laboratories, New York, New York
  - The Lipid Center, Statesville, North Carolina
  - Metabolic And Atherosclerosis Research Center, Cincinnati, Ohio
  - Sterling Research Group, Cincinnati, Ohio
  - Hospital Of The University Of Pennsylvania, Philadelphia, Pennsylvania
  - Radiant Research, Inc., Dallas, Texas
  - Baylor College Of Medicine, Houston, Texas
  - Mcallen Heart Clinic, McAllen, Texas

REFERENCES:
- [Derived] Emami H, Vucic E, Subramanian S, Abdelbaky A, Fayad ZA, Du S, Roth E, Ballantyne CM, Mohler ER, Farkouh ME, Kim J, Farmer M, Li L, Ehlgen A, Langenickel TH, Velasquez L, Hayes W, Tawakol A. The effect of BMS-582949, a P38 mitogen-activated protein kinase (P38 MAPK) inhibitor on arterial inflammation: a multicenter FDG-PET trial. Atherosclerosis. 2015 Jun;240(2):490-6. doi: 10.1016/j.atherosclerosis.2015.03.039. Epub 2015 Mar 28. PMID 25913664
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx